CLINICAL TRIAL: NCT04101981
Title: Metabolomics of Follicular Fluids in Patients Undergoing PMA
Brief Title: NMR Metabolomics Study of Follicular Fluid of Oncological Patients
Status: Completed | Type: Observational
Sponsor: San Carlo Public Hospital, Potenza, Italy (Other)
Responsible Party: Principal Investigator, Assunta Iuliano, MD, NMR metabolomics study of follicular fluid in woman with cancer resorting to fertility preservation, San Carlo Public Hospital, Potenza, Italy
Other Study IDs: NMR Metabolomics Study
Record Dates: First submitted 2018-07-27; First posted 2019-09-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Woman With Cancer Resorting Fertility Preservation
MeSH Terms: interventions — Oocyte Retrieval

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — follicular fluids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy subjects: 10 subjects
  Interventions: Procedure: oocytes retrieval
- oncological patients: 10 subjects
  Interventions: Procedure: oocytes retrieval

INTERVENTIONS:
Procedure: oocytes retrieval — The oocytes retrieval was performed after 34-36 hours from hCG administration . The collection of cumulus-oocyte complexes and FFs were performed via transvaginal ultrasound-guided aspiration with a needle of 18 gauge of diameter. The three major diameter follicles were identified by intraoperative ultrasound and FF of each follicle was collected in its own test tube.

SUMMARY:
Purpose: The purpose of this study was to evaluate the possible application of metabolomics to identify follicular fluid changes in cancer patients undergoing fertility preservation. Although metabolomics have been applied already in cancer studies, this is the first application on follicular fluid of cancer patients.

Methods: The investigators selected for the study 10 patients with breast cancer and lymphoma who resorted to oocyte cryopreservation to preserve fertility and 10 healthy women undergoing in vitro fertilization treatments. Follicular fluid was collected at the time of oocytes retrieval. Metabolomic analysis of follicular fluids was performed by 1H NMR spectroscopy in combination with multivariate analysis to interpret the spectral data. Univariate statistical analysis was applied to find correlations between patients' features and metabolites identified by NMR.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the possible application of metabolomics to identify follicular fluid changes in cancer patients undergoing fertility preservation. Although metabolomics have been applied already in cancer studies, this is the first application on follicular fluid of cancer patients.

Methods: The investigators selected for the study 10 patients with breast cancer and lymphoma who resorted to oocyte cryopreservation to preserve fertility and 10 healthy women undergoing in vitro fertilization treatments. Follicular fluid was collected at the time of oocytes retrieval. Metabolomic analysis of follicular fluids was performed by 1H NMR spectroscopy in combination with multivariate analysis to interpret the spectral data. Univariate statistical analysis was applied to find correlations between patients' features and metabolites identified by NMR.

ELIGIBILITY:
Inclusion Criteria:

* all nulliparous patients who want to have offspring, with a cancer diagnosis obtained by histological examination and with a definitive staging of the disease.

Exclusion Criteria:

* patients with suspected cancer diagnosis without histological examination and complete staging and women suffering of any cancer that received neoadjuvant chemotherapy or radiation therapy prior to follicular fluid collection.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: oncological patients with pathological diagnosis resorting fertility preservation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
follicular fluid metabolites of patients with neoplasia | NMR spectroscopy was performed immediately after oocyte retrieval
  identification by NMR spectroscopy of the metabolites present in the follicular fluid of woman

SECONDARY OUTCOMES:
to define the existence of cancer-specific metabolic profiles | NMR spectroscopy was performed immediately after oocyte retrieval
  to study by NMR spectroscopy of the existence of cancer-specific metabolic profiles present in the follicular fluid of woman resorting to fertility preservation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonietta MACM Castiglione Morelli, Professor, Principal Investigator — University of Basilicata studies; Assunta Iuliano, MD, Principal Investigator — San Carlo Public Hospital, Potenza
Locations (1):
- Angela Ostuni, Potenza, Italy

REFERENCES:
- [Background] Castiglione Morelli MA, Iuliano A, Schettini SCA, Petruzzi D, Ferri A, Colucci P, Viggiani L, Cuviello F, Ostuni A. NMR metabolomics study of follicular fluid in women with cancer resorting to fertility preservation. J Assist Reprod Genet. 2018 Nov;35(11):2063-2070. doi: 10.1007/s10815-018-1281-7. Epub 2018 Aug 1. PMID 30069850